CLINICAL TRIAL: NCT02660125
Title: Does Local Endometrial Injury Improve Implantation Rates in Women Undergoing Their First ICSI Cycle.
Brief Title: Endometrial Injury and Implantation Rates Before First ICSI Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Assistant professor, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 144
Record Dates: First submitted 2016-01-17; First posted 2016-01-21 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Invitro Fertilization
Keywords: ICSI; endometrial injury; implantation rate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endometrial scratch injury (Active Comparator): endometrial scratch done before ICSI cycle
  Interventions: Procedure: Endometrial scratch injury
- control (No Intervention): IcSI cycle without prior endometrial injury

INTERVENTIONS:
Procedure: Endometrial scratch injury — midluteal single endometrial strip will be taken using a Novak curett under general anasthesia to avoid discomfort and cramping and to proceed to cervical dilatation in case of forbidden cervix
  Arms: endometrial scratch injury

SUMMARY:
Midluteal single endometrial strip will be taken using a Novak curett under general anasthesia to avoid discomfort and cramping and to proceed to cervical dilatation in case of forbidden cervix, the step that will be beneficial to embryo transfer procedure.

Controller ovarian hyperstimulation; will be done using the long luteal phase agonist protocol and the short protocol(as judged by patient,s age ovarian reserve judged by day 3 FSH and antral follicular count and previous history of ovarian response).

Ovarian response will be monitored by vaginal ultrasound and HCG will be given when when there is >=1 follicle >=18 mm. and >=3 follicles >=16 mm. Ultasound guided oocyte retrieval will be carried out 35 hours later. Embryo transfer will be performed on day 2 or day 3 after oocyt retrieval according to number and quality of embryos.

Embryo transfer will be carried out under trans-abdominal ultrasound guidance pregnancy test will be done using qualitative blood HCG detection 2 weeks after the embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

1. subfertile women indicated for ICSI.
2. normal uterine cavity demonstrated by transvaginal ultrasound and hystrogram.
3. FSH<10mIU/mL on day 3 of her cycle.

Exclusion Criteria:

1. presence of endometrial polyp or fibroid distorting the uterine cavity.
2. hydrosalpinx.
3. ICSI carried out for preimplantation genetic diagnosis.
4. FSH>10mIU\mL.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
implantation rate | 14 days after embryo transfer
  number of sacs identifiable through ultrasonography divided by the number of embryos transferred
clinical pregnancy rate | 4 weeks after embryo transfer
  the detection of fetal cardiac activity within a gestational sac on ultrasonography examination

SECONDARY OUTCOMES:
multiple pregnancy rate | 4 weeks after embryo transfer
  number of patients who had a multifetal pregnancy divided by the total number of clinical pregnancies
abortion rate | 12 weeks of gestational age
  number of patients who had a spontaneous abortion before 12 weeks of pregnancy divided by total number of clinical pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maged AM, Rashwan H, AbdelAziz S, Ramadan W, Mostafa WAI, Metwally AA, Katta M. Randomized controlled trial of the effect of endometrial injury on implantation and clinical pregnancy rates during the first ICSI cycle. Int J Gynaecol Obstet. 2018 Feb;140(2):211-216. doi: 10.1002/ijgo.12355. Epub 2017 Nov 18. PMID 29048754